CLINICAL TRIAL: NCT00312624
Title: Morphological Predictors of Sudden Cardiac Death in Patients With Known Cardiomyopathies
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Samir Saba/Director, Cardiac electrophysiology, UPMC
Other Study IDs: 0602085; 0602085
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Cardiomyopathy
Keywords: ICD implantation; cardiac MRI; cardiomyopathy; ventricular arrhythmias; LVEF 35% or less; indication for ICD implantation as part of standard of care
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: contrast-enhanced cardiac MRI — MRI of heart with delayed enhancement

SUMMARY:
This is a pilot study to find a correlation between MRI and ICD therapy in patients with known cardiomyopathies, aiming to determine if cardiac scarring identified by MRI correlates with ventricular arrhythmias and the occurrence of ICD therapy.

DETAILED DESCRIPTION:
This is an observational study over a 3 year period of 50 patients with known cardiomyopathy and LVEF of 35% or less who will have ICD implantation as part of their standard of care. All subjects will undergo a contrast-enhanced cardiac MRI using gadolinium to determine the morphological characteristics of their left ventricle prior to ICD implant. Subjects will not be offered sedation to minimize risk, thus those suffering from claustrophobia will be excluded or dropped from participation. MRI will be evaluated, and subjects will be followed during standard of care device interrogations for 12 months after implant.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* cardiomyopathy with LVEF 35% or less
* indication for ICD implantation
* able to provide informed consent

Exclusion Criteria:

* prior device implantation
* contraindication for MRI (i.e., metallic foreign body)
* claustrophobia
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-04; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States